CLINICAL TRIAL: NCT06962527
Title: Computational Modeling of Ambiguity Aversion in Internalizing Disorders: Neural and Behavioral Markers, and a Test of Target Engagement
Brief Title: Test of Target Engagement of Ambiguity Aversion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Brent Rappaport, Assistant Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: K23MH136421 (NIH)
Record Dates: First submitted 2025-01-27; First posted 2025-05-08 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-01

CONDITIONS: Intolerance of Uncertainty; Anxiety; Intolerance of Uncertainty; Anxiety; Depression, Anxiety
Keywords: Ambiguity aversion; Intolerance of uncertainty; Computational modeling; EEG/ERP
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Participants will be aware that there is one other arm of the study to which other participants are randomized, but they will not be aware of what this other arm entails. Additionally, the intervention will be administered digitally, without a care provider, and outcome measures will be self-administered, so there is no potential for evaluator bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Uncertainty-focused single session intervention (Experimental): This is a digital, self-guided SSI that teaches adults about tolerating and embracing uncertainty in their life. The SSI is based on five elements: 1. An introduction the concept of neuroplasticity; 2. Testimonials from peers describing beliefs that people's thoughts, feelings, and behaviors are malleable, given the brain's capacity for change; 3. Strategies (from cognitive-behavioral therapy) for applying these principles to participants' lives; 4. Further vignettes by peers describing times when they tolerated or embraced uncertainty; 5. An exercise wherein participants provide advice to fictional peers, using newly-gleaned information about uncertainty,
  Interventions: Behavioral: Uncertainty-focused single session intervention
- Maintaining a healthy lifestyle single session intervention (Placebo Comparator): This is a digital, self-guided SSI that teaches adults about the benefits of maintaining a healthy lifestyle (e.g., proper sleep, diet, exercise), emphasizing recommendations by various bodies (e.g., American Medical Association). It is structurally similar to the uncertainty-focused SSI but is designed to mimic what people would receive in their annual physical with a primary care physician. The goals of this intervention is to encourage participants to identify aspects of a healthy lifestyle, and steps they could take towards a healthier lifestyle. This SSI is designed to control for nonspecific aspects of intervention, including engagement in a computer program, reading and writing exercises, and vignettes from peers.
  Interventions: Behavioral: Maintaining a healthy lifestyle single session intervention

INTERVENTIONS:
Behavioral: Uncertainty-focused single session intervention — Digitally/computer administered 30-minute self-guided intervention for adults ages 25-60
  Other Names: Uncertainty-focused SSI
  Arms: Uncertainty-focused single session intervention
Behavioral: Maintaining a healthy lifestyle single session intervention — Digitally/computer administered 30-minute self-guided intervention for adults ages 25-60
  Other Names: Maintaining a healthy lifestyle SSI
  Arms: Maintaining a healthy lifestyle single session intervention

SUMMARY:
The present work aims to test whether a single session intervention alters ambiguity aversion, both in terms of people's decision making and their brain responses to ambiguous choices.

DETAILED DESCRIPTION:
In this trial, participants will be randomized to one of two single session interventions (SSI). They will complete a decision making task before and after the SSI to measure their behavioral and brain responses to ambiguity, all on the same day. They will also complete a brief measure of hopelessness before and after the SSI. The main analysis will compare changes in ambiguity aversion before and after the interventions. Participants will also be asked to complete questionnaires before completing the task and SSI. The questionnaires will be about the participant's emotions and symptoms of depression and anxiety, personality, and avoidance/tolerance of uncertainty.

ELIGIBILITY:
Inclusion Criteria:

1. Ages 25 to 60
2. Right-handed
3. Ability to read and write English
4. Capacity to provide informed consent
5. Intolerance of uncertainty score ≥ -0.5 standard deviation below the mean (31st percentile)

Exclusion Criteria:

1. Personal history of psychosis, mania, or hypomania
2. Personal history of autism spectrum disorder
3. IQ < 80 as determined by the Wechsler Test of Adult Reading
4. Head injury with greater than 120 seconds loss of consciousness
5. Neurological condition (e.g., epilepsy, Parkinson's, cerebral palsy, history of stroke)
6. Currently pregnant
7. Use of any implanted electrical device (e.g., pacemaker, spinal stimulator, vagal nerve stimulator, Inspire sleep apnea device, etc.).

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2029-07-01 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Beck Hopelessness Scale-4 (BHS-4) | 1 hour
  The BHS-482 is a four-item self-report scale that will be used to assess hopelessness before and after the experimental intervention (scale assesses hopelessness "right now, in this moment") to determine whether the intervention was effective in eliciting change in a clinically meaningful construct. It has good psychometric properties. Participants will complete the Beck Hopelessness Scale (BHS-4) before and after the intervention as a manipulation check that the single session intervention (SSI) "worked" in the event that the other primary outcomes exhibit resistance to change.
Behavioral ambiguity aversion | 1 hour
  Computational modeling will be used to extract two parameters indicative of behavioral ambiguity aversion (AA) from a risk and ambiguity task completed once before and once after the intervention. This results in two variables per participant: one which indicates categorical AA (i.e., their tendency to choose the unambiguous choice regardless of the amount of ambiguity present) and one which indicates continuous AA (i.e., how the amount of ambiguity influences people's choice).
Event-related potential responses to ambiguous choices | 1 hour
  From EEG data collected during the risk and ambiguity task, event-related potentials (ERPs)-time-locked electroencephalogram signals with millisecond resolution-will be extracted to yield one variable per participant indicating mean brain activity to ambiguous choices. Pilot data and small prior studies have consistently found an attenuated P300-like component (albeit later than usual, around 350-500ms) to ambiguous relative to unambiguous choices similar to those on this task.

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available once they are anonymized and all the planned analyses have been completed by the investigators.
Supporting Information: SAP, Analytic Code
Time Frame: Anonymized data and code will be made publicly available upon publication of trial results, which is anticipated to be in 2030.
Access Criteria: Data will be posted of the NIMH Data Archive (NDA).